CLINICAL TRIAL: NCT02116218
Title: Assessment of Cancer Pain in Emergency Department in Traditional Chinese Medicine (TCM): A Study Protocol for a Clinical Trial
Brief Title: Assessment of Cancer Pain in Emergency Department in Traditional Chinese Medicine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated and the PI has left the institution.
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCM-2014-ED
Record Dates: First submitted 2014-04-10; First posted 2014-04-16 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Neoplasms; Pain
Keywords: Traditional Chinese Medicine; acupuncture; complementary alternative medicine; cancer pain; emergency department
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain; Emergencies | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acupuncture (Experimental): Experimental group would receive acupuncture at specific acupoints for 15 minutes.
  Interventions: Procedure: acupuncture
- seed (Sham Comparator): Control group would receive another intervention that we would put Vaccaria seeds near the acupoints but without acupressure for the same period.
  Interventions: Procedure: Vaccaria seed

INTERVENTIONS:
Procedure: acupuncture — Acupuncture in the Hegu (LI4), Shousanli (LI10), Zusanli (ST36), Yanlinquan (GB34), Taichong (LV3) and Ouch point. Needles would be correctly inserted and manually stimulated until the 'De Qi' sensation is elicited. The needles would stay in place for 15 minutes.
  Arms: acupuncture
Procedure: Vaccaria seed — We put Vaccaria seeds near the acupoints without acupressure as an intervention in control group.
  Arms: seed

SUMMARY:
Pain control is a common and serious problem in cancer patients. Although WHO has developed a three-stage model of cancer pain management, 80% cancer patients still suffer moderate to severe pain in their daily life. When patients are with acute exacerbation or aggravate of pain, they usually visit the emergency department for more help.

Acupuncture is a safe, low-invasive and economic treatment. And it has been world-wide used as a complementary therapy among patients with cancer. It can not only relieve pain in cancer patients, but also can reduce some of the side effects caused by some treatment.

This study is aimed to evaluate the efficacy and safety of acupuncture in cancer patient with acute pain onset through emergency department with objective Traditional Chinese Medicine assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 75 years, either gender.
* Visit emergency department
* Chief complaint is pain.
* Diagnosed by oncologist with International Classification of Diseases 9th revision (ICD-9) code between 140.0 to 239.9.

Exclusion Criteria:

* Serious comorbid conditions (for example, life-threatening condition).
* Patients who cannot communicate reliably with the investigator or who are not likely to obey the instructions of the trial.
* Pregnancy status.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 15 minutes after intervention
  The Visual Analog Scale (VAS) has proven its usefulness and its clinical validity for the evaluation of pain. VAS would be measured and compared before and after intervention.
Heart rate variability | 15 minutes after intervention
  Autonomic nervous dysfunction plays a role as a consequence of pain. Recording the heart rate variability (HRV) in an easy non-invasive methods to investigate autonomic balance.
  HRV would be measured and compared before and after intervention

SECONDARY OUTCOMES:
Tongue diagnosis | 15 minutes after intervention
  Tongue diagnosis plays an important role in TCM. In clinical practice Practitioners observed tongue characteristics, such as the color and shape, and the amount of saliva before deducing the primary ailment of a patient.
  We would take photos of tongue before and after intervention to compare the clinical changes.
Brief Pain Inventory | 7 days after intervention
  Brief Pain Inventory (BPI) was made by Pain Research Group in order to measure the pain score of cancer patients.
  We would do the questionnaire before and 7 days after intervention to investigate if there's a long-term effect.
adverse event | Participants will be followed for the duration of hospital stay, an expected average of 2 hours.
  Participants should report any adverse events they experience, Including discomfort or bruising at the sites of needle insertion, nausea, or feeling faint after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lun-Chien Lo, Study Chair — Changhua Christian Hospital
Locations (1):
- Changhua Christian hospital, Changhua, Taiwan

REFERENCES:
- [Background] Garcia MK, McQuade J, Haddad R, Patel S, Lee R, Yang P, Palmer JL, Cohen L. Systematic review of acupuncture in cancer care: a synthesis of the evidence. J Clin Oncol. 2013 Mar 1;31(7):952-60. doi: 10.1200/JCO.2012.43.5818. Epub 2013 Jan 22. PMID 23341529
- [Background] Chiu J, Yau T, Epstein RJ. Complications of traditional Chinese/herbal medicines (TCM)--a guide for perplexed oncologists and other cancer caregivers. Support Care Cancer. 2009 Mar;17(3):231-40. doi: 10.1007/s00520-008-0526-x. Epub 2008 Nov 14. PMID 19009311
- [Background] van den Beuken-van Everdingen MH, de Rijke JM, Kessels AG, Schouten HC, van Kleef M, Patijn J. Prevalence of pain in patients with cancer: a systematic review of the past 40 years. Ann Oncol. 2007 Sep;18(9):1437-49. doi: 10.1093/annonc/mdm056. Epub 2007 Mar 12. PMID 17355955
- [Background] Azevedo Sao Leao Ferreira K, Kimura M, Jacobsen Teixeira M. The WHO analgesic ladder for cancer pain control, twenty years of use. How much pain relief does one get from using it? Support Care Cancer. 2006 Nov;14(11):1086-93. doi: 10.1007/s00520-006-0086-x. Epub 2006 Jun 8. PMID 16761128